Statistical Analysis: Data was analyzed by using SPSS Statistics for Windows, Version 23.0 (IBM SPSS Statistics for Windows, Version 23.0. Armonk, NY: IBM Corp). Descriptive data was compared using Chi-Square and Mann-Whitney U tests, while Wilcoxon's and McNemar's tests were used to compare the menstruation findings of the students before and after the training. Dependent Samples t-Test was used in the intragroup comparison of total HLBS-II, MSQ, and sub-dimension scores. Comparison of differences between groups was performed by using the Independent Samples t-Test. Pearson's correlation analysis was used to determine the relationship between total HLBS-II and MSQ scores.